CLINICAL TRIAL: NCT05837156
Title: A Multicenter, Randomized, Single-blind, Parallel Controlled Clinical Study of Cyclopofol Injection for the Prevention of Postoperative Nausea and Vomiting
Brief Title: A Clinical Study to Evaluate Cyclopofol Injection for the Prevention of Postoperative Nausea and Vomiting
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mengchang Yang (Other)
Responsible Party: Sponsor-Investigator, Mengchang Yang, Deputy Chief Physician, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 950429
Record Dates: First submitted 2023-04-02; First posted 2023-05-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Nausea and Vomiting
Keywords: Cyclophenol; Heptaflurane
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group cyclophenol (Active Comparator): Calculated by body weight (kg), the initial dose of continuous infusion of cyclopophenol is 0.8 mg/kg/h. During the infusion, the researchers adjusted the rate according to the reaction of the subjects, and the adjustment range was 0.4 mg/kg/h-2.4 mg/kg/h.
  Interventions: Drug: Cyclophenol
- group heptaflurane (Active Comparator): The anesthetic sevoflurane is inhaled for anesthesia maintenance. The initial concentration of sevoflurane is 1.5-2.0%, which can be adjusted to the expected effect according to the subject's reaction.
  Interventions: Drug: Heptaflurane
- group heptaflurane combined cyclophenol (Experimental): Inhaled anesthetic sevoflurane combined with a small dose of cyclopophenol for anesthesia maintenance. The initial concentration of sevoflurane is 0.5%, and the initial dose of cyclopophenol is 0.4 mg/kg/h.After that, sevoflurane or cyclopophenol (with an adjustment range of 0.2 mg/kg/h-1.2 mg/kg/h) can be adjusted to the expected effect according to the subject's reaction.
  Interventions: Drug: Heptaflurane combined Cyclophenol

INTERVENTIONS:
Drug: Heptaflurane combined Cyclophenol — Heptaflurane combined Cyclophenol
  Arms: group heptaflurane combined cyclophenol
Drug: Heptaflurane — Heptaflurane only
  Arms: group heptaflurane
Drug: Cyclophenol — Cyclophenol only
  Arms: group cyclophenol

SUMMARY:
This study uses cyclopropofol as a positive control and adopts a large sample, multicenter, randomized, single-blind, positive parallel control test design to explore the clinical application value of cyclopropofol in preventing postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Before the end of the anesthesia maintenance period/operation, it was divided into groups A, B and C according to different drug regimens. The subjects were randomly assigned to one of them in a 1:1:1 ratio to receive cyclopophenol or sevoflurane anesthesia. Each group of subjects should be roughly consistent according to the proportion of each number of PO . After screening the object, the researchers of each testing center are confirmed by the researchers of the center, log in to the random system, fill in the screening information, obtain the random number information, and distribute the corresponding research drugs according to the random number. The number of random shelters is generated through SAS software, which is used as a centralized random grouping system to import the total number of drugs. This study sets up evaluation researchers and drug management researchers. The whole experimental process turned a blind eye to not only the subjects, but also the evaluators. This study has set up evaluation investigators and administrative investigators. Administrative researchers are only involved in the random grouping, dispensing and delivery process. Other processes, including the subject's informed consent, screening, efficacy indicators and safety evaluation, and planned visits, are completed by the evaluation investigators.

ELIGIBILITY:
Inclusion Criteria:

1. At least 2 of the 4 induced risk factors of PONV (risk factors are: history of PONV or motion sickness, habitual non-smoking, women, receiving opioid analgesia).
2. For patients with an estimated duration of anesthesia ≥1h and ≤3h (non-emergency, non-cardiothoracic surgery and non-intracranial surgery), laparoscopic surgery, gastrointestinal surgery, obstetrics and gynecology surgery, tympanoplasty, tonstonectomy, etc., are preferred. The duration of hand anesthesia was defined as the period from the beginning of anesthesia induction to the end of anesthesia maintenance
3. Male or female, age ≥ 18 years old, ASA-PS score I to III.

Exclusion Criteria:

1. There is a history of vestibular nerve disorder or dizziness or nausea and vomiting 24 hours before the operation; or receiving conventional antiemetic treatment.
2. The subjects who need to maintain ventilation after surgery or need to place the nasogastric tube in place for a period of time.
3. The subject who the researcher believes that there are any other factors that are not suitable to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-08-02 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of PONV within 24 hours after each group's operation. | Day 1
  PONV incidence (%) = (number of patients with nausea and vomiting / number of PONV incidence (%) = (number of patients with nausea and vomiting / number of people in the group) × 100%

SECONDARY OUTCOMES:
The incidence of nausea and vomiting within 48 hours after surgery in each group | Day 2
  PONV incidence (%) = (number of patients with nausea and vomiting / number of PONV incidence (%) = (number of patients with nausea and vomiting / number of people in the group) × 100%
The average number of rescues within 24 and 48 hours after surgery in each group | Day 2
  Severe vomiting (level 3 or above) requires rescue treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Sichuan, China

IPD SHARING:
Plan to Share IPD: No